CLINICAL TRIAL: NCT00609544
Title: A Multi-Center, Double-Blind, Placebo-Controlled Safety and Preliminary Efficacy Study of IL-1 Trap (Rilonacept) Administered Subcutaneously in Subjects With Non Dialysis-Dependent Chronic Kidney Disease (NDD-CKD) and Anemia
Brief Title: Study of the Safety and Effectiveness of Rilonacept (IL-1 Trap) Administered Subcutaneously in Subjects With Non Dialysis-Dependent Chronic Kidney Disease (NDD-CKD) and Anemia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to enroll patients
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Gary Swergold MD, PhD / Medical Director, Regeneron Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IL1T-AN-0704
Record Dates: First submitted 2007-12-10; First posted 2008-02-07 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Chronic Kidney Disease; Anemia
Keywords: Non Dialysis-dependent chronic kidney disease and anemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia | interventions — rilonacept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Rilonacept
- 2 (Placebo Comparator)
  Interventions: Drug: Rilonacept

INTERVENTIONS:
Drug: Rilonacept — Loading dose of 320 mg Rilonacept or placebo followed by 160 mg Rilonacept or placebo once a week for 11 weeks

SUMMARY:
Anemia of inflammation is a common complication in patients with chronic kidney disease (CKD). Patients with CKD and anemia of inflammation also exhibit decreased response to erythropoietic agents, even in the presence of adequate iron stores. This decreased responsiveness is associated with increased levels of proinflammatory cytokines. Rilonacept is being developed for the treatment of inflammatory disorders.

This is a clinical research study to determine the safety and effectiveness of rilonacept for the treatment of anemia in inflamed patients with CKD who are not yet on dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female greater than 18 years of age
* Chronic Kidney Disease (CKD) not yet requiring renal replacement therapy (pre-dialysis patients)
* Not expected to require dialysis during duration of the study
* Adequate laboratory values
* If on rHuEPO therapy, the dose must be stable

Exclusion Criteria:

* Persistent chronic or active infections
* Intravenous (IV) iron administration within 12 weeks prior to the Screening Visit
* Known history of severe uncontrolled hyperparathyroidism
* Prior recipient or scheduled to receive a kidney transplant during the study
* Abnormal laboratory values
* Unstable angina or myocardial infarction within the past 6 months prior to the Screening Visit
* Uncontrolled hypertension
* Coronary disease diagnosed in the 3 months prior to the Screening Visit
* Severe Congestive Heart Failure
* History of HIV
* Hepatitis B and/or Hepatitis C
* Abnormal chest radiograph
* A positive intradermal skin tuberculin test
* History or presence of cancer within 5 years of the Screening Visit
* History of alcohol abuse or current intake of 21 or more alcohol-containing drinks per week
* History of drug abuse within the 5 years prior to the Screening Visit
* Lactating females or pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Change in blood hemoglobin concentration. | Baseline to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Gary Swergold, MD, PhD, Study Director — Regeneron Pharmaceuticals
Locations (27):
- United States (27):
  - Alexander City, Alabama
  - Muscle Shoals, Alabama
  - Cerritos, California
  - Long Beach, California
  - Los Alampios, California
  - Thousand Palms, California
  - Colorado Springs, Colorado
  - Lauderdale Lakes, Florida
  - Pembroke Pines, Florida
  - Tampa, Florida
  - Blue Ridge, Georgia
  - Jonesboro, Georgia
  - Portland, Maine
  - Queens, New York
  - Mooresville, North Carolina
  - Shelby, North Carolina
  - Allentown, Pennsylvania
  - Harrisburg, Pennsylvania
  - Orangeburg, South Carolina
  - Sumter, South Carolina
  - Barlett, Tennessee
  - Clarksville, Tennessee
  - Collierville, Tennessee
  - Crossville, Tennessee
  - Memphis, Tennessee
  - Ogden, Utah
  - Falls Church, Virginia